CLINICAL TRIAL: NCT06496555
Title: Evaluation of U-AKIpredTM for Predicting AKI in Critically Ill Patients Within 12 Hours: a Multicenter Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, tao zhihua, Professor, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2024-0605
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: External Effectiveness Validation of Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of our study is to evaluate U-AKIpredTM for predicting AKI in critically ill patients within 12 h by the multicenter prospective cohorts. AKI was diagnosed by Kidney Disease Improving Global Outcomes (KDIGO) criteria. We designed five aspects including the overall fitting effecience evaluation, calibration curve, quantifying calibration performance, quantifying discrimination performance, quantifying clinical utility to evaluate the external validation model.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients who stayed in ICU for over 24 h;
* patients older than 18 years of age.

Exclusion Criteria:

* patients who admitted in ICU had been diagnosed acute kidney injury;
* patients who admitted in ICU had been diagnosed acute kidney disease;
* patients who admitted in ICU had been diagnosed chronic kidney disease;
* patients who admitted in ICU had performed kidney dialysis;
* patients who admitted in ICU had performed kidney transplantation;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Probability Sample
Enrollment: 2100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AKI occurrence | 12 hours

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China